CLINICAL TRIAL: NCT05673408
Title: Non-Invasive Blood Pressure Validation Study
Brief Title: NIBP Validation Study
Status: Recruiting | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: CC_MA_NIBPValidation_2022_1151
Record Dates: First submitted 2023-01-03; First posted 2023-01-06 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness
Keywords: NIBP Validation; Non-Invasive Blood Pressure
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Subject Group 1: Neonates, Infant, Children <3 years of age
  Interventions: Device: Philips IntelliVue X3 Patient Monitor
- Subject Group 2: Children 3-12 years of age
  Interventions: Device: Philips IntelliVue X3 Patient Monitor
- Subject Group 3: Adolescent/Adult >12 years of age
  Interventions: Device: Philips IntelliVue X3 Patient Monitor

INTERVENTIONS:
Device: Philips IntelliVue X3 Patient Monitor — All subjects enrolled in this study will receive one Philips non-invasive blood pressure cuff. This cuff will be connected via compatible hose to the Philips IntelliVue X3 monitor hosting the released or investigational NIBP algorithm. The invasive blood pressure from the radial arterial line will also be connected to the Philips IntelliVue X3 monitor. The Philips IntelliVue X3 monitor will in turn be connected to a laptop for data collection.

SUMMARY:
The purpose of this study is to compare measurements of blood pressure (BP) between the Philips non-invasive blood pressure (NIBP) system (including NIBP cuff and portable patient monitor) and invasive radial for Subject Group 2 and 3, and radial or umbilical arterial line for neonates (A-line) in critical care patients.

DETAILED DESCRIPTION:
A multi-center, multi-phase, prospective, self-controlled, observational study.

* Phase I - A pilot phase designed for feasibility and the potential for algorithm development (enhancement).
* Phase II - Pivotal Phase: At the completion of Phase I -and finalization of the algorithm (if applicable), Phase II is designed for the purpose of establishing equivalence of the Philips NIBP system with the gold standard radial or umbilical (neonates) arterial line.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted into the NICU, PICU, ICU, or OR (operating room)
* Adult aged 18 years and older, or parent/legal guardian of minor, willing and able to understand and provide informed consent/assent
* Indication for NIBP cuff
* Indication for radial arterial line for Subject Group 2 and Subject Group 3, and radial or umbilical arterial line for Subject Group 1
* Meet the following stratification criteria across the study:

Stratification (per the ISO 81060-2:2018/Amd-2:2024):

* Subject Group 1:

  * At least 3 patients shall be <1000 g in weight
  * At least 3 patients shall be 1000 to 2000 g in weight
  * At least 3 patients shall be > 2000 g in weight
  * At least 3 patients shall be ≥ 29 days and < 1 year of age
  * At least 3 patients shall be ≥ 1 year and < 3 years of age
  * The remaining patients may be from any of the above age or weight groups in order to complete the sample size
  * A patient can be in more than one category simultaneously
* Subject Group 2:

  * At least 30% male, 30% female
  * Limb circumference distributed as specified in ISO81060-2:2018/Amd2:2024.
* Subject Group 3:

  * At least 30% male, 30% female
  * Limb circumference distributed as specified in ISO81060- 2:2018/Amd-2:2024.
  * At least 10% SBP ≤ 100mmHg
  * At least 10% SBP ≥ 160mmHg
  * At least 10% DBP ≤ 70mmHg
  * At least 10% DBP ≥ 85mmHg

Exclusion Criteria:

* Inability to place the study device appropriately due to patient's anatomy or condition
* Known pregnancy or lactating women (self-report)
* Patients treated with an intra-aortic balloon pump
* Aortic and mitral regurgitation (> 2 nd degree)
* Measurements taken in the lateral position
* Currently participating in another clinical trial with any product, treatment and/or medication that clinically interferes with the study endpoint(s)
* If valid SBP reference measurements for lateral difference is > 15 mmHg (except for neonates with umbilical A-line)
* If valid DBP reference measurements for lateral difference is > 10 mmHg (except for neonates with umbilical A-line)
* At the Principal Investigator's discretion, subject does not qualify to participate in the study for any reasons that are not mentioned above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The clinical study will be conducted in neonate, infant, pediatric, and adult patients admitted into the NICU/PICU/ICU/OR.
Sampling Method: Probability Sample
Enrollment: 189 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Philips NIBP System Equivalence to Radial Arterial Line | Through study completion, approximately 1 year
  The primary endpoint is the accuracy and precision of systolic blood pressure (SBP), diastolic blood pressure (DBP), and mean arterial pressure (MAP) measured by the Philips NIBP system (including NIBP cuff and portable patient monitor) in comparison to radial arterial line.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - University Health Women's and Children's Hospital, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided